CLINICAL TRIAL: NCT04184362
Title: Empower Opioid Misuse Theranova Study for Veterans With Chronic Pain
Brief Title: Empower Opioid Misuse & Chronic Pain
Acronym: RAP_EOM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-27491
Record Dates: First submitted 2019-10-23; First posted 2019-12-03 (Actual); Results first posted 2023-08-03 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-07

CONDITIONS: Chronic Pain; Opioid Use
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Experimental group tested at the active treatment site (Experimental): The theranova empower device will be tested at the active treatment site.
  Interventions: Device: Empower Neuromodulation System Transcutaneous Electrical Nerve Stimulation
- Control sham group tested at the sham control treatment site (Sham Comparator): The theranova empower device will be tested the sham control treatment site.
  Interventions: Device: Empower Neuromodulation System Transcutaneous Electrical Nerve Stimulation

INTERVENTIONS:
Device: Empower Neuromodulation System Transcutaneous Electrical Nerve Stimulation — Participants will self-administer treatment with the Empower device two times daily for two weeks. Participants will complete surveys over the two-week period to evaluate the effects of the Empower treatment.

SUMMARY:
This study evaluates the effects of peripheral nerve stimulation on opioid craving and use and pain in participants with chronic non-cancer pain (NCP) and opioid misuse. Participants will be randomized to receive the active or sham control treatment for the duration of the study.

DETAILED DESCRIPTION:
This pilot study aims to examine the feasibility, acceptability, and preliminarily examine efficacy of peripheral nerve stimulation with the Empower Neuromodulation System on reducing opioid craving and use and decreasing pain. Opioid prescribing for chronic pain has increased dramatically over the past several decades, with devastating public health consequences, including high rates of opioid misuse and overdose deaths. Safe nonpharmacological treatments are urgently needed. In this randomized, controlled study, thirty Veterans with chronic non-cancer pain (NCP) and opioid misuse will be recruited and randomly assigned (1:1) to either the Active or Control treatment. On Days 1-7, participants will undergo baseline monitoring, and on Days 8-21, participants will undergo daily nerve stimulation treatment. Pain scores, craving, and opioid use will be measured daily Days 0-21. Our goal is to provide an intervention that, alone or in conjunction with current treatments, reduces craving and reduces reliance on opioids in high-risk chronic pain patients.

ELIGIBILITY:
Inclusion Criteria:

* VA-eligible Veterans
* Ages 18-75
* Currently prescribed and taking chronic opioids (≥90 days dispensed in past 12 months) for non-malignant, non-palliative pain
* Current (past 12 months) opioid misuse, defined as opioid use not as prescribed. Participants with COMM ≥ 9, SOAPP-R ≥ 18, and/or medical and pharmacy records reflective of opioid misuse in the past 12 months.

Exclusion Criteria:

* Injury or damage to the ulnar nerve, and/or neuropathy in the upper extremities
* Pregnant or planning to become pregnant
* Currently implanted with an electrical and/or neurostimulator device, including cardiac pacemaker or defibrillator, vagal neuro-stimulator, deep brain stimulator, spinal stimulator, sacral stimulator, bone growth stimulator, or cochlear implant
* Use of an investigational drug/device therapy within the past 4 weeks
* Current medical or psychiatric instability as determined by the participant's primary care provider and/or study PI
* Severe opioid use disorder (OUD) requiring medication-assisted therapy (buprenorphine, methadone, or naltrexone IM) for OUD
* Injury or nerve damage at the arm or palm that prevents safe use of Empower device at either site
* Unable to provide informed written consent
* Prone to epilepsy or seizures

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-11-20 (Actual); Primary Completion 2022-03-21 (Actual); Study Completion 2022-03-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Herbst, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- San Francisco VA Medical Center, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 245 potentials received outreach materials. 204 potentials connected with the study staff. 115 potentials consented for pre-screening.
Period: Overall Study
Arm/Group | Experimental Group Tested at the Active Treatment Site | Control Sham Group Tested at the Sham Control Treatment Site
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental Group Tested at the Active Treatment Site | Control Sham Group Tested at the Sham Control Treatment Site | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 2 | 2
  >=65 years | 5 | 3 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 70 (4.6) | 64 (13) | 67 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 4 | 5 | 9
Race/Ethnicity, Customized [Number; unit: participants]
  Race: White | 3 | 5 | 8
  Race: Black or African American | 1 | 0 | 1
  Race: Unknown or Not Reported | 1 | 0 | 1
  Ethnicity: Unknown or Not Reported | 1 | 0 | 1
  Ethnicity: Not Hispanic or Latino | 4 | 5 | 9
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Pain Intensity Score Measures
Description: Each participant will be given the Empower app and trained on app use. They will record pain levels daily on the Empower app, with a 0-100 scale. 0 indicating a lack of pain outcome, and 100 indicating maximum pain score. Pain score measures will be taken throughout the study. The Empower App will prompt all participants daily to complete the Numeric Rating Scale to assess pain levels immediately before and after treatment.
  Participants complete daily measures of Visual Analog Scale for scores on Numeric Rating Pain Scale, to assess pain intensity before and after treatment or sham condition. The data reported is the mean average of all scores taken daily from baseline to week 3, and reflects scores from both before and after treatment.
Time Frame: Baseline to Week 3
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Experimental Group Tested at the Active Treatment Site | Control Sham Group Tested at the Sham Control Treatment Site
Number analyzed (Participants) | 5 | 5
Score on a scale | 55 (25) | 57 (22)

2. Primary Outcome: Opioid Craving Intensity With Empower Neuromodulation Active Treatment Versus Control Treatment
Description: Each participant will be given the Empower app and trained on app use. They will record craving levels daily on the Empower app, with a 0-100 scale. 0 indicating an outcome with a lack of craving, and 100 indicating an outcome with maximum craving intensity.
  The Empower App will prompt all participants daily to complete the following measure of Visual Analog Scale, to assess craving intensity before and after treatment.
  Participants complete daily measures of Visual Analog Scale, to assess craving immediately before and after treatment or sham condition. The data reported is the mean average of all scores taken daily from baseline to week 3, and reflects scores from both before and after treatment.
Time Frame: Baseline to Week 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Group Tested at the Active Treatment Site | Control Sham Group Tested at the Sham Control Treatment Site
Number analyzed (Participants) | 5 | 5
score on a scale | 29 (20) | 33 (35)

3. Primary Outcome: Mean Morphine Equivalent Doses: Opioid Use With Empower Active Treatment Versus Control Treatment
Description: The Empower App will prompt all participants daily to complete the measure of prescribed and nonprescribed self-reported opioid use for the previous day, and morphine equivalents will be recorded weekly through timeline follow back reviews with staff.
  Population being treated at active and sham sites report opioid use, in Morphine Equivalent (mg) doses.
Time Frame: Baseline to Week 3
Measure: Mean (Standard Deviation); unit: Morphine Equivalents (mg)
Arm/Group | Experimental Group Tested at the Active Treatment Site | Control Sham Group Tested at the Sham Control Treatment Site
Number analyzed (Participants) | 5 | 5
Morphine Equivalents (mg) | 1882 (3040) | 336 (387)

4. Secondary Outcome: General Health Monitored
Description: General health measures will be monitored through surveys administered through Qualtrics (except for Week 0 screening visit surveys). The surveys will be emailed to participants to measure multidimensional assessment of interoceptive awareness (MAIA-2) 0-5 scale, physical activity (PAS-2) records average activity time per week, brief anxiety inventory (BAI) 0-3 scale, insomnia severity index (ISI) with a 0-4 scale, and distress intolerance index (DII) with a 0-4 scale. Increased MAIA-2 & PAS2, or decreased BAI, ISI, and DII show improvement.
Time Frame: Treatment Time Frame: Week 1 to Week 3
Population: Data for this outcome measure were not collected and therefore can not be reported here.
Arm/Group | Experimental Group Tested at the Active Treatment Site | Control Sham Group Tested at the Sham Control Treatment Site
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 weeks
Arm/Group | Experimental Group Tested at the Active Treatment Site | Control Sham Group Tested at the Sham Control Treatment Site
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5

LIMITATIONS AND CAVEATS:
We enrolled our first 5 participants before March 2020. During March 2020, the UCSF and SFVAHCS Research Offices announced that all non-essential in-person clinical activities had to be suspended effective immediately due to the COVID-19 pandemic and shelter-in-place order in the San Francisco Bay Area. In 2021, we received IRB approval to conduct remote study visits. This older population with chronic pain also faced a lot of technical issues, dealing with virtual meetings and measures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-01): https://cdn.clinicaltrials.gov/large-docs/62/NCT04184362/Prot_SAP_001.pdf